CLINICAL TRIAL: NCT04300751
Title: Interactions of Alcohol and Opioids: Pharmacodynamic Effects
Brief Title: The Behavioral Effects of Opioids and Alcohol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sharon Walsh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Walsh, Director of the Center on Drug and Alcohol Research, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 55176; R01DA016718 (NIH)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use; Alcohol Drinking
Keywords: opioid; opiate; alcohol
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a randomized, double-blind, double-dummy, placebo-controlled, within-subjects design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alcohol (Experimental): Participants will receive experimental doses of active or placebo alcohol, p.o. Alcohol/placebo will be administered once per session.
  Interventions: Drug: Alcohol
- Opioid Agonist (Experimental): Participants will receive non-therapeutic, experimental doses of an active opioid agonist or placebo. Active opioid agonist/placebo will be administered once per session and will be administered orally
  Interventions: Drug: Opioid Agonist
- Opioid Agonist/Alcohol Combination (Experimental): Participants will receive non-therapeutic, experimental doses of active opioid/placebo in combination with experimental doses of active alcohol placebo. Opioid/placebo and alcohol/placebo doses will be administered once during each session. It is possible to receive both active drugs on the same day. Both opioid and alcohol doses will be administered orally.
  Interventions: Drug: Alcohol; Drug: Opioid Agonist

INTERVENTIONS:
Drug: Alcohol — Active alcohol or placebo, administered orally
  Arms: Alcohol; Opioid Agonist/Alcohol Combination
Drug: Opioid Agonist — Active opioid agonist or placebo, administered orally
  Arms: Opioid Agonist; Opioid Agonist/Alcohol Combination

SUMMARY:
This study will examine the effects of doses of alcohol/placebo and doses of opioid/placebo, alone and in combination. The primary outcomes are related to pharmacodynamic measures (subjective ratings of drug liking and other abuse-related effects; physiological outcomes) to determine the interaction effects of these compounds.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 21-55
* Current non-medical use of opioids
* Previous alcohol use

Exclusion Criteria:

* Physical dependence on opioids, alcohol, or benzodiazepines/sedative/hypnotics
* Seeking treatment for drug use
* Significant medical problems

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Walsh, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover study with 9 conditions tested in random order in each completing subject.
Groups:
- The Behavioral Effects of Opioids and Alcohol: Participants will receive non-therapeutic, experimental doses of active opioid/placebo in combination with experimental doses of active alcohol placebo. Opioid/placebo and alcohol/placebo doses will be administered once during each session. It is possible to receive both active drugs on the same day. Both opioid and alcohol doses will be administered orally.
  Alcohol: Active alcohol or placebo, administered orally
  Opioid Agonist: Active opioid agonist or placebo, administered orally
Period: Overall Study
Arm/Group | The Behavioral Effects of Opioids and Alcohol
Started | 11
Placebo/Placebo | 10
Oxycodone 20mg/Placebo | 10
Oxycodone 40mg/Placebo | 10
Placebo/Alcohol 0.5g/kg | 10
Placebo/Alcohol 0.8g/kg | 11
Oxycodone 20mg/Alcohol 0.5g/kg | 10
Oxycodone 20mg/Alcohol 0.8g/kg | 10
Oxycodone 40mg/Alcohol 0.5g/kg | 11
Oxycodone 40mg/Alcohol 0.8g/kg | 10
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One participant did not complete the study. They left the study for non-study related reasons.
Groups:
- Alcohol and Opioids: Participants will receive non-therapeutic, experimental doses of active opioid/placebo in combination with experimental doses of active alcohol placebo. Opioid/placebo and alcohol/placebo doses will be administered once during each session. It is possible to receive both active drugs on the same day. Both opioid and alcohol doses will be administered orally.
  Alcohol: Active alcohol or placebo, administered orally
  Opioid Agonist: Active opioid agonist or placebo, administered orally
Arm/Group | Alcohol and Opioids
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.30 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Peak Subject-Rated Outcome: Visual Analog Scale (VAS) Drug Liking
Description: Participants rated their subjective drug liking on a standardized VAS scale (0 to 100; 0=Not at all, 100=Extremely). A higher score indicates greater drug liking. This outcome was recorded multiple times at regular intervals throughout the experimental dose condition sessions. For each dose condition, the participants' peak value was pulled from the raw data and averaged to yield one mean (SEM).
Time Frame: These outcomes (visual analog scores, scale of 0-100) are recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session)
Population: Per Protocol population, defined as participants completing the 9 experimental dosing conditions.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo/Placebo; Oxycodone 20mg/Placebo; Oxycodone 40mg/Placebo; Placebo/Alcohol 0.5g/kg; Placebo/Alcohol 0.8g/kg; Oxycodone 20mg/Alcohol 0.5g/kg; Oxycodone 20mg/Alcohol 0.8g/kg; Oxycodone 40mg/Alcohol 0.5g/kg; Oxycodone 40mg/Alcohol 0.8g/kg: Participants will receive non-therapeutic, experimental doses of active opioid/placebo in combination with experimental doses of active alcohol/placebo. Opioid/placebo and alcohol/placebo doses will be administered once during each session. It is possible to receive both active drugs on the same day. Both opioid and alcohol doses will be administered orally.
  Alcohol: Active alcohol or placebo, administered orally
  Opioid Agonist: Active opioid agonist or placebo, administered orally
Arm/Group | Placebo/Placebo | Oxycodone 20mg/Placebo | Oxycodone 40mg/Placebo | Placebo/Alcohol 0.5g/kg | Placebo/Alcohol 0.8g/kg | Oxycodone 20mg/Alcohol 0.5g/kg | Oxycodone 20mg/Alcohol 0.8g/kg | Oxycodone 40mg/Alcohol 0.5g/kg | Oxycodone 40mg/Alcohol 0.8g/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
score on a scale | 12.9 (8.6) | 47.1 (9.4) | 49.9 (7.9) | 54.8 (8.8) | 61.2 (8.2) | 54.6 (9.4) | 66.9 (9.4) | 57.2 (9.1) | 72.9 (7.2)

2. Secondary Outcome: Peak Subject-Rated Outcome: Visual Analog Scale (VAS) - How Drunk do You Feel?
Description: Participants rated their subjective response to the question "How drunk do you feel?" on a standardized VAS scale (0 to 100; 0=Not at all, 100=Extremely). A higher score indicates greater feeling of drunk. TThis outcome was recorded multiple times at regular intervals throughout the experimental dose condition sessions. For each dose condition, the participants' peak value was pulled from the raw data and averaged to yield one mean (SEM).
Time Frame: as for outcome 1
Population: Per Protocol population, defined as participants completing the 9 experimental dosing conditions.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo/Placebo | Oxycodone 20mg/Placebo | Oxycodone 40mg/Placebo | Placebo/Alcohol 0.5g/kg | Placebo/Alcohol 0.8g/kg | Oxycodone 20mg/Alcohol 0.5g/kg | Oxycodone 20mg/Alcohol 0.8g/kg | Oxycodone 40mg/Alcohol 0.5g/kg | Oxycodone 40mg/Alcohol 0.8g/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
score on a scale | 6.1 (4.7) | 6.5 (5.7) | 8.6 (5.0) | 41.2 (7.6) | 54 (7.6) | 39.6 (8.3) | 49.5 (8.5) | 33.4 (8.2) | 56.1 (8.7)

3. Secondary Outcome: Trough Oxygen Saturation
Description: Oxygen saturation (measured as a percentage through pulse ox) monitored throughout each session. Lower scores indicate greater impairment. This outcome was recorded multiple times at regular intervals throughout the experimental dose condition sessions. For each dose condition, the participants' trough value was pulled from the raw data and averaged to yield one mean (SEM).
Time Frame: Oxygen Saturation recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: Percentage of oxygen in blood
Arm/Group | Placebo/Placebo | Oxycodone 20mg/Placebo | Oxycodone 40mg/Placebo | Placebo/Alcohol 0.5g/kg | Placebo/Alcohol 0.8g/kg | Oxycodone 20mg/Alcohol 0.5g/kg | Oxycodone 20mg/Alcohol 0.8g/kg | Oxycodone 40mg/Alcohol 0.5g/kg | Oxycodone 40mg/Alcohol 0.8g/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Percentage of oxygen in blood | 97.4 (0.35) | 96.8 (0.29) | 96.6 (0.36) | 96.6 (0.43) | 96.2 (0.30) | 96.1 (0.34) | 95.7 (0.30) | 95.6 (0.49) | 95.2 (0.47)

4. Secondary Outcome: Peak Cold Pressor Test Threshold
Description: Participants immerse their forearm in cold water (1.0 +/- .5 degree Celsius) and remove their arm from the cold water to indicated pain tolerance (max 5 mins). Cold Pressor Test Threshold (time elapsed since cold water immersion measured in seconds) monitored throughout each session. Higher scores indicate greater impairment. This outcome was recorded multiple times at regular intervals throughout the experimental dose condition sessions. For each dose condition, the participants' peak value was pulled from the raw data and averaged to yield one mean (SEM).
Time Frame: Cold Pressor Test Threshold was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo/Placebo | Oxycodone 20mg/Placebo | Oxycodone 40mg/Placebo | Placebo/Alcohol 0.5g/kg | Placebo/Alcohol 0.8g/kg | Oxycodone 20mg/Alcohol 0.5g/kg | Oxycodone 20mg/Alcohol 0.8g/kg | Oxycodone 40mg/Alcohol 0.5g/kg | Oxycodone 40mg/Alcohol 0.8g/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Seconds | 22.6 (7.3) | 63.3 (30.2) | 74.2 (32.4) | 43.4 (24.2) | 60.6 (31.7) | 54.1 (20.1) | 73.2 (31.9) | 81.5 (30.0) | 98.9 (30.9)

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks. Adverse Event (AE) monitoring begins once consent is signed and is tracked through participant disqualification or follow-up visit.
Description: AE definitions are the same as the clnicaltrials.gov definitions.
Groups:
- Pre-Intervention / Days Off: Prior to any drug administration or on participant days off when AE is not related to drug conditions.
- Qualification: Oxycodone 30mg / Placebo: Prior to the experimental conditions, participants will receive a non-therapeutic dose of oxycodone 30 mg, p.o. during a qualifying day session. This session serves as a responsive challenge which is intended to confirm that subjects are able to detect the active drug.
Arm/Group | Pre-Intervention / Days Off | Qualification: Oxycodone 30mg / Placebo | Placebo/Placebo | Oxycodone 20mg/Placebo | Oxycodone 40mg/Placebo | Placebo/Alcohol 0.5g/kg | Placebo/Alcohol 0.8g/kg | Oxycodone 20mg/Alcohol 0.5g/kg | Oxycodone 20mg/Alcohol 0.8g/kg | Oxycodone 40mg/Alcohol 0.5g/kg | Oxycodone 40mg/Alcohol 0.8g/kg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/11 | 2/11 | 1/10 | 0/11 | 1/10 | 1/10 | 1/10 | 0/10 | 0/11 | 0/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Intervention / Days Off (N=11) | Qualification: Oxycodone 30mg / Placebo (N=11) | Placebo/Placebo (N=10) | Oxycodone 20mg/Placebo (N=11) | Oxycodone 40mg/Placebo (N=10) | Placebo/Alcohol 0.5g/kg (N=10) | Placebo/Alcohol 0.8g/kg (N=10) | Oxycodone 20mg/Alcohol 0.5g/kg (N=10) | Oxycodone 20mg/Alcohol 0.8g/kg (N=11) | Oxycodone 40mg/Alcohol 0.5g/kg (N=10) | Oxycodone 40mg/Alcohol 0.8g/kg (N=10)
Diarrrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized Body Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea / Vomitting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT04300751/Prot_SAP_ICF_001.pdf